CLINICAL TRIAL: NCT07224737
Title: Machine Learning-based Exosome Liquid Biopsy Enables Stratification of Occult Metastasis Risk in Patients With Intrahepatic Cholangiocarcinoma
Brief Title: Liquid Biopsy Using Exosomal miRNA Enables Risk Stratification of Potential Metastasis in Patients With Intrahepatic Cholangiocarcinoma.
Acronym: EXOMIC
Status: Recruiting | Type: Observational
Sponsor: City of Hope Medical Center (Other)
Responsible Party: Sponsor
Other Study IDs: 23228/EXOMIC
Record Dates: First submitted 2025-11-03; First posted 2025-11-05 (Actual); Last update posted 2025-11-10 (Actual); Status verified 2025-11

CONDITIONS: Intrahepatic Cholangiocarcinoma (Icc)
Keywords: Exosomal miRNA; ICC; Liquid Biopsy; Occult metastasis; Tumor recurrence; Liver cancer
MeSH Terms: conditions — Cholangiocarcinoma; Cirrhosis, Familial, with Pulmonary Hypertension; Recurrence; Liver Neoplasms

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (6):
- Training Cohort - ICC with Occult Metastasis: The cohort of ICC patients who had occult metastasis detected at the time of surgery.
  Preoperative samples were analyzed using the EXOMIC qRT-PCR assay to validate candidate exosomal microRNAs identified in the discovery cohort.
  Interventions: Diagnostic Test: EXOMIC assay (qRT-PCR validation)
- Training Cohort - ICC without Occult Metastasis: The cohort of ICC patients without occult metastasis at the time of surgery. Preoperative samples were analyzed with the EXOMIC qRT-PCR assay to evaluate differential miRNA expression and refine the predictive model for occult metastasis detection.
  Interventions: Diagnostic Test: EXOMIC assay (qRT-PCR validation)
- Validation Cohort - ICC with Occult Metastasis: The cohort of ICC patients with occult metastasis at the time of primary tumor resection.
  The EXOMIC qRT-PCR assay was applied to confirm the predictive value of the exosomal miRNA panel in identifying occult metastasis prior to surgery.
  Interventions: Diagnostic Test: EXOMIC assay (qRT-PCR validation)
- Validation Cohort - ICC without Occult Metastasis: The cohort of ICC patients without occult metastasis at the time of surgery. Preoperative samples were analyzed with the EXOMIC qRT-PCR assay to evaluate differential miRNA expression and refine the predictive model for occult metastasis detection.
  Interventions: Diagnostic Test: EXOMIC assay (qRT-PCR validation)
- Discovery Cohort - ICC with Occult Metastasis: Patients with intrahepatic cholangiocarcinoma (ICC) who were found to have occult metastasis at the time of primary tumor resection in the discovery cohort.
  Preoperative samples were analyzed using small RNA sequencing to identify exosome-derived microRNAs associated with the presence of occult metastasis.
  Interventions: Diagnostic Test: EXOMIC small RNA sequencing
- Discovery Cohort - ICC without Occult Metastasis: Patients with ICC who had no occult metastasis at the time of primary tumor resection in the discovery cohort.
  Preoperative samples from these patients were analyzed by small RNA sequencing and compared with those from patients with occult metastasis to identify candidate microRNAs.
  Interventions: Diagnostic Test: EXOMIC small RNA sequencing

INTERVENTIONS:
Diagnostic Test: EXOMIC small RNA sequencing — High-throughput small RNA sequencing performed on preoperative serum or plasma samples from patients with intrahepatic cholangiocarcinoma (ICC) to identify exosome-derived microRNAs associated with occult metastasis at the time of surgery.
  Sequencing data were analyzed to detect differentially expressed miRNAs between patients with and without occult metastasis in the discovery cohort.
  Groups: Discovery Cohort - ICC with Occult Metastasis; Discovery Cohort - ICC without Occult Metastasis
Diagnostic Test: EXOMIC assay (qRT-PCR validation) — Quantitative reverse transcription PCR (qRT-PCR)-based validation of candidate exosomal microRNAs identified through small RNA sequencing.
  This assay was performed on preoperative serum or plasma samples from independent ICC patient cohorts to validate the predictive value of selected miRNAs for occult metastasis detection prior to surgical resection.
  Groups: Training Cohort - ICC with Occult Metastasis; Training Cohort - ICC without Occult Metastasis; Validation Cohort - ICC with Occult Metastasis; Validation Cohort - ICC without Occult Metastasis

SUMMARY:
Occult metastasis at the time of surgery is a major driver of poor outcomes in intrahepatic cholangiocarcinoma (ICC), yet reliable preoperative biomarkers to identify such patients are lacking. The EXOMIC study aims to develop and validate a circulating exosomal microRNA (exo-miRNA)-based liquid biopsy assay to detect occult metastasis preoperatively in patients with resectable ICC.

DETAILED DESCRIPTION:
Intrahepatic cholangiocarcinoma (ICC) incidence is rising globally, and prognosis remains poor. Patients harboring occult micrometastases that are not detected on preoperative imaging often experience rapid recurrence and significantly worse survival. Tumor-derived exosomes contribute to pre-metastatic niche formation and carry microRNAs that reflect aggressive metastatic potential. Circulating exosomal microRNA profiles may serve as non-invasive biomarkers to reveal occult metastasis before surgery.

Preoperative exosomes will be analyzed using small RNA sequencing (discovery) followed by RT-qPCR validation and machine-learning modeling to develop a predictive score for occult metastasis. The study will evaluate diagnostic performance (sensitivity, specificity, accuracy, AUROC), prognostic relevance (OS/RFS), and clinical utility (decision curve analysis) to establish a biologically informed framework for treatment stratification in ICC.

ELIGIBILITY:
Inclusion Criteria:

* Histologically confirmed ICC (clinical stage I-III).
* Undergoing curative-intent hepatectomy.
* Availability of preoperative pasma or serum sample (≥200 µL).
* Standard staging imaging completed per institutional protocol.
* Written informed consent.

Exclusion Criteria:

* Extrahepatic cholangiocarcinoma or gallbladder cancer.
* Synchronous non-ICC malignancy.
* Inadequate clinical follow-up.
* Inability to consent.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: 250
Sampling Method: Non-Probability Sample
Enrollment: 250 (Estimated)
Dates: Start 2024-06-21 (Actual); Primary Completion 2026-06-18 (Estimated); Study Completion 2026-06-18 (Estimated)

PRIMARY OUTCOMES:
Recurrence Free Survival | 3 years
  The time period from surgery to recurrence of ICC.

SECONDARY OUTCOMES:
Overall Survival | 5 years
  Time from surgery to death from any cause

CONTACTS AND LOCATIONS:
Overall Officials: Ajay Goel, PhD, Principal Investigator — City of Hope Medical Center
Locations (1):
- City of Hope Medical Center, Duarte, California, United States

IPD SHARING:
Plan to Share IPD: No
Data collected for the study will be made available to others, including de-identified participant data, at publication, via a signed data access agreement and at the discretion of the investigators' approval of the proposed use of such data.

REFERENCES:
- [Background] Huang G, Zhang H, Yang Z, Li Q, Yuan H, Chen P, Xie C, Meng B, Zhang X, Chen K, Yu H. Predictive value of HTS grade in patients with intrahepatic cholangiocarcinoma undergoing radical resection: a multicenter study from China. World J Surg Oncol. 2024 Jan 11;22(1):17. doi: 10.1186/s12957-023-03281-6. PMID 38200585
- [Background] Swanson K, Wu E, Zhang A, Alizadeh AA, Zou J. From patterns to patients: Advances in clinical machine learning for cancer diagnosis, prognosis, and treatment. Cell. 2023 Apr 13;186(8):1772-1791. doi: 10.1016/j.cell.2023.01.035. Epub 2023 Mar 10. PMID 36905928
- [Background] Kojima T, Umeda Y, Fuji T, Niguma T, Sato D, Endo Y, Sui K, Inagaki M, Oishi M, Ota T, Hioki K, Matsuda T, Aoki H, Hirai R, Kimura M, Yagi T, Fujiwara T. Efficacy of surgical management for recurrent intrahepatic cholangiocarcinoma: A multi-institutional study by the Okayama Study Group of HBP surgery. PLoS One. 2020 Sep 3;15(9):e0238392. doi: 10.1371/journal.pone.0238392. eCollection 2020. PMID 32881910
- [Background] Feng J, Liang B, Zhang HY, Liu Z, Jiang K, Zhao XQ. Prognostic factors for patients with mass-forming intrahepatic cholangiocarcinoma: A case series of 68 patients. World J Gastrointest Surg. 2022 May 27;14(5):442-451. doi: 10.4240/wjgs.v14.i5.442. PMID 35734620
- [Background] Doussot A, Gonen M, Wiggers JK, Groot-Koerkamp B, DeMatteo RP, Fuks D, Allen PJ, Farges O, Kingham TP, Regimbeau JM, D'Angelica MI, Azoulay D, Jarnagin WR. Recurrence Patterns and Disease-Free Survival after Resection of Intrahepatic Cholangiocarcinoma: Preoperative and Postoperative Prognostic Models. J Am Coll Surg. 2016 Sep;223(3):493-505.e2. doi: 10.1016/j.jamcollsurg.2016.05.019. Epub 2016 Jun 11. PMID 27296525
- [Background] Yu TH, Chen X, Zhang XH, Zhang EC, Sun CX. Clinicopathological characteristics and prognostic factors for intrahepatic cholangiocarcinoma: a population-based study. Sci Rep. 2021 Feb 17;11(1):3990. doi: 10.1038/s41598-021-83149-5. PMID 33597569
- [Background] Clements O, Eliahoo J, Kim JU, Taylor-Robinson SD, Khan SA. Risk factors for intrahepatic and extrahepatic cholangiocarcinoma: A systematic review and meta-analysis. J Hepatol. 2020 Jan;72(1):95-103. doi: 10.1016/j.jhep.2019.09.007. Epub 2019 Sep 16. PMID 31536748
- [Background] Bertuccio P, Malvezzi M, Carioli G, Hashim D, Boffetta P, El-Serag HB, La Vecchia C, Negri E. Global trends in mortality from intrahepatic and extrahepatic cholangiocarcinoma. J Hepatol. 2019 Jul;71(1):104-114. doi: 10.1016/j.jhep.2019.03.013. Epub 2019 Mar 23. PMID 30910538
- [Background] An L, Zheng R, Zhang S, Chen R, Wang S, Sun K, Lu L, Zhang X, Zhao H, Zeng H, Wei W, He J. Hepatocellular carcinoma and intrahepatic cholangiocarcinoma incidence between 2006 and 2015 in China: estimates based on data from 188 population-based cancer registries. Hepatobiliary Surg Nutr. 2023 Feb 28;12(1):45-55. doi: 10.21037/hbsn-21-75. Epub 2021 Jul 21. PMID 36860251
- [Background] Sirica AE, Strazzabosco M, Cadamuro M. Intrahepatic cholangiocarcinoma: Morpho-molecular pathology, tumor reactive microenvironment, and malignant progression. Adv Cancer Res. 2021;149:321-387. doi: 10.1016/bs.acr.2020.10.005. Epub 2020 Dec 9. PMID 33579427
- [Background] Fiste O, Ntanasis-Stathopoulos I, Gavriatopoulou M, Liontos M, Koutsoukos K, Dimopoulos MA, Zagouri F. The Emerging Role of Immunotherapy in Intrahepatic Cholangiocarcinoma. Vaccines (Basel). 2021 Apr 22;9(5):422. doi: 10.3390/vaccines9050422. PMID 33922362
- [Background] Zhang R, Wang Z, Yang M, Chen B, Liu M, Zheng M, Liu PX, Wang L. Combining traditional analysis and machine learning to predict early, middle, and long-term recurrence of intrahepatic cholangiocarcinoma. Eur J Surg Oncol. 2025 Sep;51(9):110141. doi: 10.1016/j.ejso.2025.110141. Epub 2025 May 9. PMID 40446770
- [Background] Zhao B, Cheng Q, Cao H, Zhou X, Li T, Dong L, Wang W. Dynamic change of serum CA19-9 levels in benign and malignant patients with obstructive jaundice after biliary drainage and new correction formulas. BMC Cancer. 2021 May 7;21(1):517. doi: 10.1186/s12885-021-08204-w. PMID 33962560